CLINICAL TRIAL: NCT03950193
Title: Association Between Presence and Parental Participation in Perinatal Care and Child Psychiatric Profile at 24 Months After Preterm Birth
Brief Title: Prematurity and Parental Involvement in Child Development Care
Acronym: parentpart
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19055
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Premature Birth
Keywords: Parental presence; parental involvement; parental stress; development care; psychic development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premature child: Premature children evaluated during their 24 months follow up consultation
  Interventions: Other: Questionnaires to evaluate psychic development of the child

INTERVENTIONS:
Other: Questionnaires to evaluate psychic development of the child — Child Behaviour Checklist. This test, completed by parents and with 52 questions, is designed to screen children at high risk for emotional problems, mood disorders, anxiety, pervasive developmental problems, attention deficit and hyperactivity, antonymic reactions (oppostion, provocation) and sleep problems.

SUMMARY:
The aims of the study is to evaluate the association between presence and parental participation in perinatal care and psychic development of the child at 24 months

DETAILED DESCRIPTION:
In France, as in developed countries, the premature birth rate has been rising over the past few years. Premature labor is a particularly stressful birth. It is recognized that the level of parental stress is greater at a premature birth compared to a term birth. The neuro-developmental consequences of premature birth are important. A possible association between prematurity and the onset of mental disorders such as hyperactivity, inattention, emotional problems, conduct disorders, autistic disorders and social difficulties has been shown. It has been shown that parental presence, holding and skin to skin during hospitalization would be beneficial for the child's motor development and psychological well-being by reducing the stress of the child.

ELIGIBILITY:
inclusion criteria : child born very prematurely between 27 and 31 weeks gestational age + 6 days child taken in charge at the intensive care unit of Reims University Hospital for at least 3 weeks child aged 24 months (+/- 2 months) the holders of parental authority are more 18 years old the holders of parental authority know how to speak, read and write French the holders of parental authority agree to participate in the study

exclusion criteria :

- child has a serious pathology (abnormal brain MRI)

Ages: 22 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premature children
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Child Behavior Check List | Day 0
  This test, completed by parents and with 52 questions, is designed to screen children at high risk for emotional problems, mood disorders, anxiety, pervasive developmental problems, attention deficit and hyperactivity, antonymic reactions (oppostion, provocation) and sleep problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France